CLINICAL TRIAL: NCT02126787
Title: Short-term, Intensive Psychodynamic Group Therapy Versus Cognitive-behavioral Group Therapy in the Day Treatment of Anxiety Disorders and Comorbid Depressive or Personality Disorders
Brief Title: Short-term, Intensive Psychodynamic Group Therapy Versus Cognitive-behavioral Group Therapy in the Day Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Wola Hospital (Unknown); University of Warsaw (Other)
Responsible Party: Principal Investigator, Andrzej Kokoszka, Professor, MD, PhD, Medical University of Warsaw
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NN402464340
Record Dates: First submitted 2014-04-09; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Anxiety Disorders; Depressive Disorders; Personality Disorders
Keywords: Anxiety disorders; Depressive disorders; Personality disorders; Psychodynamic psychotherapy; Cognitive-behavioral psychotherapy; Group psychotherapy; Day treatment
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Personality Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intensive Group Analytic Psychotherapy (Experimental): Intensive Group Analytic Psychotherapy in a day clinic setting
  Interventions: Behavioral: Intensive Group Analytic Psychotherapy
- Intensive GCBT (Experimental): Intensive transdiagnostic cognitive-behavioral group therapy in a day clinic setting
  Interventions: Behavioral: Intensive transdiagnostic cognitive-behavioral group therapy
- Wait-list control group (No Intervention)

INTERVENTIONS:
Behavioral: Intensive Group Analytic Psychotherapy — The form of intensive group analytic therapy to be used in the trial has been manualized by the research team for the study. It is rooted in group analysis tradition (Bion 1961; Foulkes & Anthony, 1965). It is based on two recent group analytic psychotherapy manuals, one developed by Lorentzen (2014), the other by Garland (2010). The manual has been adapted to day treatment setting and also draws on polish psychoanalytical group experiences practiced in a public service. Like in other psychodynamic short-term therapies this approach is more structured and focused on issues relevant to symptoms relief. Thereby additional techniques are used: psychodrama, non-verbal techniques, movie therapy, memoir, summary or relaxation.
  Arms: Intensive Group Analytic Psychotherapy
Behavioral: Intensive transdiagnostic cognitive-behavioral group therapy — GCBT was designed for treatment in naturalistic settings of diagnostically mixed anxiety disorder patients with comorbid Personality Disorders (PD's) (Holas, Szaniawska, Suszek, Błażejewski, & Kokoszka, in prep.). It is based on the transdiagnostic approach to emotional and particularly anxiety disorders that has been developed over the past ten years (Barlow, 2000; Barlow, Allen, & Choate, 2004; Norton, 2006), additionally it includes interventions for personality disorders based of schema therapy and modes of personality disorders. This approach assumes a high overlap between anxiety disorders and is focused on the common aspects of them. Intensive GCBT developed by our group shares the classical assumptions of cognitive-behavioral therapy (Beck, 1976).
  Arms: Intensive GCBT

SUMMARY:
Background: Psychodynamic and cognitive-behavioral group therapies are frequently applied in day hospitals in the treatment of anxiety disorders, and comorbid depressive or personality disorders in Poland. There is not enough evidence for its effectiveness in this environment. This study addresses this gap. The aim is to determine the effectiveness of the two kinds of day treatments consisting of intensive, short-term group therapy: psychodynamic and cognitive-behavioral for patients with anxiety disorders and comorbid depressive or personality disorders. Our objectives are: 1) Demonstrating effectiveness of each treatment in a day care setting relative to wait-list control; 2) Demonstrating the relative short- and long-term effectiveness of the two active treatments; 3) Preliminary examination of predictors and moderators of treatment response; and 4) Preliminary examination of mediators of therapeutic change; 5) Detailed comparison of impact of both methods of treatment on the outcome of used measures.

Methods/design: In this randomized controlled trial, a total of 123 patients with anxiety disorders and comorbid depressive or personality disorders will be assigned to one of three conditions: 1) psychodynamic group therapy; 2) cognitive-behavioral group therapy; 3) waiting list (control group). Therapy will last 12 weeks. Both treatments will be manualized (manuals will address comorbidity). Primary outcome measures are include self-report symptoms of anxiety, observer rated symptoms of anxiety, global improvement and dichotomized diagnosis of anxiety disorder. Secondary outcome measures include personality, depression, self-esteem, defense mechanisms, beliefs about self and others, interpersonal problems, object relations, parental bonding, meta-cognition, mindfulness and quality of life: symptoms of anxiety, depression, personality, self-esteem and defense mechanisms. Measures are taken at baseline, post-treatment and 3 months following the end of the therapy.

Discussion: The randomized controlled trial format is used to compare effectiveness of intensive group cognitive-behavior therapy and intensive group psychodynamic therapy for anxiety disorders and comorbid depressive or personality disorders. The rationale is to investigate how effectively anxiety disorders and comorbid personality disorders can be treated in a day hospital typical for Polish healthcare system in 3 months treatment.

DETAILED DESCRIPTION:
Anxiety disorders are among the most prevalent mental disorders, with lifetime prevalence of 30% in US (Kessler et al., 2005) and only 9,9% in Poland (Moskalewicz, Wciórka, Kiejna, Wojtyniak, 2012), the study of the similar methodology, like in the U.S. Many studies suggest their strong comorbidity with personality disorders in some countries. Recent meta-analysis of 125 studies conducted by Friborg, Martinussen, Kaiser, Overgård and Rosenvinge (2013) has shown that a risk of comorbid anxiety disorders and personality disorders varies from 35% to 52%. Alongside anxiety disorders, the most frequently co-occurring are cluster C personality disorders. Epidemiologic studies also show high comorbidity rates for anxiety and depressive disorders, ranging from 40%-80% (Jacobi et al., 2004; Lamers et al., 2011). The data on relationships between comorbid mental disorders and treatment outcome is inconsistent. Reviews by Reich and Green (1991) and Reich and Vasile (1993) including 38 studies have shown that comorbid anxiety disorders and personality disorders are negatively related to treatment outcome. However, Dressen and Arntz (1997) after analyzing 15 studies do not share these conclusions.

Day treatment care is directed precisely to the patients who need treatment of a greater intensity and cannot be treated in outpatient care. Group psychotherapy (often used together with pharmacotherapy) is employed in day care since the 1940s (cf. Cameron 1947; Goldman, 1989). This form of therapy is chosen on economic basis. The treatment usually takes place a few days a week and lasts for several months. Different types of psychotherapy or different treatment methods (e.g. therapeutic community, psychodrama, art therapy, psycho-drawing, movie therapy, social skills training) are often applied together. In Poland, group psychotherapy is widely used in day care. Nowadays 300 such wards exist in Poland. Psychotherapy for anxiety disorders and personality disorders lasting for few months (most often three months) is provided for approximately 8000 patients a year (IPIN, 2009).

The effectiveness of day care is investigated to a very small degree, compared to its frequent usage (cf. Marshall et al 2001). However, difficulties in identifying the basic effective components of the treatment and a large diversity of treatment programs make it difficult to generalize the results.

Among a scarce number of published studies, only four were randomized controlled trials (RCT). Three of these studies compared psychotherapy in day care units to outpatient psychotherapy (Tyler et al., 1987; Dick et al., 1991; Arnevik et al., 2009) and one study used a waiting list control group (Piper, Rosie, Azim, & Joyce, 1993). Tyler et al. (1987) found no significant differences between day care and outpatient care for anxiety disorders. Dick et al. (1991) found a significant difference in the improvement of personality disorder pathology, in favor of day care. In the first study psychotherapy modality was not mentioned, in the second an eclectic psychotherapy was applied. In another study Arnevik et al. (2009), day care (18 week group psychodynamic and cognitive-behavioral psychotherapy) was compared to individual psychotherapy in patients with personality disorders and no significant differences in improvement were observed between the two groups. Piper et al. (1993) found that day care patients suffering from affective disorders and personality disorders experienced a significant improvement that continued in follow-up after 8 months (18 week group psychodynamic psychotherapy), compared to patients in a waiting list control group. Authors of a Cochrane review of day care versus outpatient care notice that because of a small number of existing studies: "there is only limited evidence to justify the provision of day treatment programs and transitional day hospital care, and no evidence to support the provision of day care centers" (Marshall et al. 2001). Existing data is therefore not sufficient to justify the use of group psychotherapy in day care, and more high quality research is needed. The question of which treatment of the two most widely used, psychodynamic or CBT, is more effective also awaits an answer. These questions are relevant in light of the large expenditures incurred by the national health funds financing the treatment. They are also important for the health care in Poland, where this type of treatment is very common.

Objectives

The main objective of the planned research is to evaluate the clinical effectiveness of intensive, short-term, psychodynamic and cognitive-behavioral group psychotherapy for an anxiety disorders with comorbid depressive or personality disorders in day care conditions.

More specific objectives are: 1) Demonstrating effectiveness of each treatment in a day care setting relative to wait-list control; 2) Demonstrating the relative short- and long-term effectiveness of the two active treatments; 3) Preliminary examination of predictors and moderators of treatment response; and 4) Preliminary examination of mediators of therapeutic change; 5) Detailed comparison of impact of both methods of treatment on the outcome of used measures.

Study design

This study is a randomized controlled trial (RCT) in which participants will be allocated to one of the three conditions: 1) psychodynamic group therapy; 2) cognitive-behavioral group therapy; 3) or a waiting-list control group (WL). Participants allocated to the waiting list condition start their treatment after 12-week waiting period. The total duration of the study will be three years. Figure 1 shows the trial design. The study protocol, information brochure and informed consent were approved by the Medical Ethics Committee of the Warsaw Medical University.

Study center

The protocol and the design is part of the research grant given to the II Department of Psychiatry Medical University of Warsaw. The study will be carried out at the day unit Wola Center of Mental Health at Hospital of Wola in Warsaw that is used as clinical setting of the II Department of Psychiatry Medical University of Warsaw.

Participants (recruitment, inclusion and exclusion criteria, randomization)

Participants with anxiety disorders and comorbid personality disorders will be recruited in outpatient clinic. Subjects who meet all the inclusion criteria will be randomized to two modalities of treatments and the waiting list. Inclusion and exclusion criteria are listed in Table 1. The number of excluded patients and reasons for exclusion will be recorded. The diagnostic criteria are based on the DSM-V system. Independent researchers not involved in the treatment will make diagnosis of personality with with the Structured Clinical Interview for DSM-IV Axis II Disorders (SCID-II; First, Gibbon, Spitzer, Williams, Benjamin, 1997, 2010) and of clinical disorders with International Neuropsychiatric Interview 5 (M.I.N.I.; Sheehan et al., 1998; Masiak & Przychoda, 1998). Diagnosis and qualification to treatment modality is carried out during ambulatory sessions. Up to 6 individual sessions will be required for the recruitment procedure including 3 sessions with a certified clinical psychologist, 2 sessions with a psychiatrist, and one for outcome measures. Pharmacological consultation take place before randomization. Waiting time before admission is planned to be between 4 and 8 weeks. Participants will be randomized using random numbers tables. Baseline measurement will occur a day before the beginning of therapy. A recruitment flow chart is presented in Figure 1. Patients are planned to be enrolled in the study over a period of three years. Before participating in the study, each patient will be provided with written information about the study and invited to give written consent for inclusion. Participants who will not meet the inclusion criteria will be offered suitable alternative treatment options. The focus of the treatment is on psychotherapy, but a medication is continued or initiated if necessary during the screening procedure at least 4 weeks before the beginning of a group psychotherapy (stable medical treatments with SSRI or SNRI without dose changes during psychotherapy). Due to high comorbidity of anxiety and depressive disorders, depressive disorders patients with mild depression disorders were not excluded, however patients with main depressive pathology were not included.

Assessments

Patients are subjected to 4 assessments: 1) at screening; 2) baseline after randomization; 3) in the end of the 12 weeks treatment; 4) six months after the end of the therapy, in order to evaluate longer-term effects of the treatments. Information from the screening is used to perform stratified randomization and to validate inclusion and exclusion criteria. Patients are assessed by independent and trained clinicians, who are blind to treatment conditions and who will not be involved in the direct clinical care of any of them. Primary outcome measures and secondary outcome measures can be distinguished in this study. Primary outcome measures include self-report symptoms of anxiety, observer rated symptoms of anxiety, global improvement and dichotomized diagnosis of anxiety disorder. Secondary outcome measures include personality, depression, self-esteem, defense mechanisms, beliefs about self and others, interpersonal problems, object relations, parental bonding, meta-cognition, mindfulness and quality of life. The following socio-demographic data will be collected: sex, age, marital status, education, past treatments, symptom history, medication. We also examine patients' expectancy for change and treatment. Some of the variables (e.g. presence or absence of a personality disorder) will be treated in exploratory analyses as predictors and moderators of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Axis I anxiety disorder (based on M.I.N.I.)
* Diagnosis of comorbid personality disorder (based on SCID II) or depressive disorder (based on M.I.N.I.)
* Age: 18 to 65 years
* Sufficient knowledge of the Polish language
* Written informed consent of the patient

Exclusion Criteria:

* Organic disorder
* Acute substance related disorders
* Schizophrenia, bipolar affective disorder
* Severe depression [over 26 points in Beck Questionnaire] or bipolar disorder.
* Dissocial personality disorder, schizotypal personality disorder
* Current suicidal ideation with a high risk of suicide
* Restriction of intellectual capacity
* Serious unstable medical problems/complications
* Concurrent psychotherapeutic treatment
* Failed treatment of CBT or psychodynamic psychotherapy for anxiety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory | week 0 (baseline)
  State-Trait Anxiety Inventory (STAI; Spielberger, Gorsuch, Lushene, Vagg, Jacobs, 1983; Polish version: Wrześniewski, Sosnowski, Matusik, 2002). The STAI measures a person's situational (or state) anxiety, as well as the amount of anxiety a person generally feels most of the time (trait). The two self-report scales contain 20 items each.
Hamilton Anxiety Rating Scale | week 0 (baseline)
  Hamilton Anxiety Rating Scale (HAM-A; Hamilton, 1959; Polish translation). The HAM-A is an interviewer-administered and rated measure of the severity of anxiety symptoms. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety).
Clinical Global Impression - Severity scale | week 0 (baseline)
  Clinical Global Impression - Severity scale (CGI-S; Guy, 1976; Polish translation). CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
Clinical Global Impression - Improvement scale | week 0 (baseline)
  Clinical Global Impression - Improvement scale (CGI-I; Guy, 1976; Polish translation). CGI-I is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Mini-International Neuropsychiatric Interview 5 | week 0 (screening)
  Mini-International Neuropsychiatric Interview 5 (M.I.N.I.; Sheehan et al., 1998; Polish version: Masiak & Przychoda, 1998). M.I.N.I. is a short diagnostic interview based on the DSM-IV criteria that focus on the existence of current psychiatric disorders. It consists of separate modules to diagnose specific disorders.
Becks Depression Inventory II | week 0 (screening)
  Becks Depression Inventory II (BDI-II; Beck, Brown & Steer, 1996; Polish version: Zawadzki, Popiel & Pragłowska, 2009) is a 21-item self-report inventory used to assess DSM-IV depressive symptoms. Each item consists of four statements, indicating increasing symptom severity.
State-Trait Anxiety Inventory | week 12 (end of treatment)
  State-Trait Anxiety Inventory (STAI; Spielberger, Gorsuch, Lushene, Vagg, Jacobs, 1983; Polish version: Wrześniewski, Sosnowski, Matusik, 2002). The STAI measures a person's situational (or state) anxiety, as well as the amount of anxiety a person generally feels most of the time (trait). The two self-report scales contain 20 items each.
Hamilton Anxiety Rating Scale | week 12 (end of treatment)
  Hamilton Anxiety Rating Scale (HAM-A; Hamilton, 1959; Polish translation). The HAM-A is an interviewer-administered and rated measure of the severity of anxiety symptoms. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety).
Clinical Global Impression - Severity scale | week 12 (end of treatment)
  Clinical Global Impression - Severity scale (CGI-S; Guy, 1976; Polish translation). CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
Clinical Global Impression - Improvement scale | week 12 (end of treatment)
  Clinical Global Impression - Improvement scale (CGI-I; Guy, 1976; Polish translation). CGI-I is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Mini-International Neuropsychiatric Interview 5 | week 12 (end of treatment)
  Mini-International Neuropsychiatric Interview 5 (M.I.N.I.; Sheehan et al., 1998; Polish version: Masiak & Przychoda, 1998). M.I.N.I. is a short diagnostic interview based on the DSM-IV criteria that focus on the existence of current psychiatric disorders. It consists of separate modules to diagnose specific disorders.
Becks Depression Inventory II | week 12 (end of treatment)
  Becks Depression Inventory II (BDI-II; Beck, Brown & Steer, 1996; Polish version: Zawadzki, Popiel & Pragłowska, 2009) is a 21-item self-report inventory used to assess DSM-IV depressive symptoms. Each item consists of four statements, indicating increasing symptom severity.
State-Trait Anxiety Inventory | week 24 (follow-up)
  State-Trait Anxiety Inventory (STAI; Spielberger, Gorsuch, Lushene, Vagg, Jacobs, 1983; Polish version: Wrześniewski, Sosnowski, Matusik, 2002). The STAI measures a person's situational (or state) anxiety, as well as the amount of anxiety a person generally feels most of the time (trait). The two self-report scales contain 20 items each.
Hamilton Anxiety Rating Scale | week 24 (follow-up)
  Hamilton Anxiety Rating Scale (HAM-A; Hamilton, 1959; Polish translation). The HAM-A is an interviewer-administered and rated measure of the severity of anxiety symptoms. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety).
Clinical Global Impression - Severity scale | week 24 (follow-up)
  Clinical Global Impression - Severity scale (CGI-S; Guy, 1976; Polish translation). CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
Clinical Global Impression - Improvement scale | week 24 (follow-up)
  Clinical Global Impression - Improvement scale (CGI-I; Guy, 1976; Polish translation). CGI-I is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Mini-International Neuropsychiatric Interview 5 | week 24 (follow-up)
  Mini-International Neuropsychiatric Interview 5 (M.I.N.I.; Sheehan et al., 1998; Polish version: Masiak & Przychoda, 1998). M.I.N.I. is a short diagnostic interview based on the DSM-IV criteria that focus on the existence of current psychiatric disorders. It consists of separate modules to diagnose specific disorders.
Becks Depression Inventory II | week 24 (follow-up)
  Becks Depression Inventory II (BDI-II; Beck, Brown & Steer, 1996; Polish version: Zawadzki, Popiel & Pragłowska, 2009) is a 21-item self-report inventory used to assess DSM-IV depressive symptoms. Each item consists of four statements, indicating increasing symptom severity.

SECONDARY OUTCOMES:
Structured Clinical Interview for DSM-IV Personality Disorders Questionnaire | week 0 (screening)
  Structured Clinical Interview for DSM-IV Personality Disorders Questionnaire (SCID-II; First et al., 1997, Polish version: First et al., 2010). SCID-II is an observer-based diagnostic interview used to determine DSM-IV Axis II disorders.
Symptoms Checklist | week 0 (baseline)
  Symptoms Checklist (SCL-90-R; Derogatis, 1994; Polish translation). SCL-90-R consists of 90 items and is designed to evaluate a broad range of psychological problems and symptoms of psychopathology. It measures 9 primary symptom dimensions and is designed to provide an overview of a patient's symptoms and their intensity at a specific point in time.
Self-Esteem Scale | week 0 (baseline)
  Self-Esteem Scale (SES; Rosenberg, 1965; Polish version: Dzwonkowska, Lachowicz-Tabaczek & Łaguna, 2008). The SES is a 10-item self-report scale that measures global self-worth by measuring both positive and negative feelings about the self.
Defense Style Questionnaire | week 0 (baseline)
  Defense Style Questionnaire (DSQ-40; Andrews, Singh & Bond M, 1993; Polish version: Bogutyn, Kokoszka, Pałczyński & Holas, 1999). The DSQ-40 is a 40 item self-report questionnaire designed to measure an individual's propensity towards three various defense styles (mature, neurotic and immature) along with twenty individual defense mechanisms.
Personality Beliefs Questionnaire | week 0 (baseline)
  Personality Beliefs Questionnaire (PBQ; Beck & Beck, 1991; Polish translation). The PBQ is a 126-item self-report measure of beliefs associated with 10 DSM-III-R and DSM-IV personality disorders (represented as subscales): 1) avoidant; 2) dependent; 3) obsessive-compulsive; 4) histrionic; 5) passive-aggressive; 6) narcissistic; 7) paranoid; 8) schizoid; 9) antisocial, and 10) borderline.
Inventory of Interpersonal Problems | week 0 (baseline)
  Inventory of Interpersonal Problems (IIP; Horowitz, Alden, Wiggins, & Pincus 2000; Polish translation). The IIP is a 64-item self-report questionnaire that inventories the interpersonal problems that people experience. It contains eight scales that assess different aspects of an individual's interpersonal difficulties: 1) domineering/controlling; 2) vindictive/self-centered; 3) cold/distant; 4) socially inhibited; 5) non-assertive; 6) overly accommodating; 7) self-sacrificing; 8) intrusive/needy.
Dysfunctional Working Models Scale | week 0 (baseline)
  Dysfunctional Working Models Scale (DWM-S; Perris, Fowler, Skagerlind, Olsson & Thorsson, 1998; Polish version: Nieznański, Habrat, Szyszkowski, Chojnowska & Walczak, 2001). The DWM-S is a 35-item self-report measure of dysfunctional working models of self and others.
Experiences in Close Relationships | week 0 (baseline)
  Experiences in Close Relationships (ECR; Brennan , Clark & Shaver, 1998; Polish version: Stawska, 2010). The ECR is a 36-item self-report measure of adult attachment. It groups people into four different categories on the basis of scores along two scales: avoidance and anxiety.
Bell Object Relations and Reality Testing Inventory | week 0 (baseline)
  Bell Object Relations and Reality Testing Inventory (BORRTI; Bell, 1995; Polish version: Staniszewski, 2011). The BORRTI is a 45-item self-report measure designed to evaluate the ability to sustain essential relationships and accurately identify internal and external reality.
Meta-cognitions Questionnaire | week 0 (baseline)
  Meta-cognitions Questionnaire (MCQ; Cartwright-Hatton & Wells, 1997; Polish version: Gawęda & Kokoszka, 2013). The MCQ is a 65-item self-report scale developed to assess several dimensions of metacognition thought to be relevant to psychopathology. Its ﬁve subscales are: 1) positive beliefs about worry; 2) negative beliefs about thoughts concerning uncontrollability and danger; 3) cognitive conﬁdence (assessing conﬁdence in attention and memory); 4) negative beliefs concerning the consequences of not controlling thoughts, and 5) cognitive self-consciousness (the tendency to focus attention on thought processes).
Five Facet Mindfulness Questionnaire | week 0 (baseline)
  Five Facet Mindfulness Questionnaire (FFMQ-S; Baer et al. 2006; Polish translation). FFMQ-S is a 39-item self-report measure which assesses five facets of a general tendency to be mindful in daily life: observing, describing, acting with awareness, nonreactivity to inner experience, and nonjudging of inner experience.
Satisfaction With Life Scale | week 0 (baseline)
  Satisfaction With Life Scale (SWLS; Diener, Emmons, Larsen & Griffin, 1985; Polish version: Juczyński, 2001). The SWLS is a 5-item self-report global measure of life satisfaction.
Credibility/Expectancy Questionnaire | week 0 (baseline)
  Credibility/Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000; Polish translation). CEQ is used to measure expectancy for change and treatment credibility as potential confounds for outcome. It comprises six questions.
Symptoms Checklist | week 12 (end of treatment)
  Symptoms Checklist (SCL-90-R; Derogatis, 1994; Polish translation). SCL-90-R consists of 90 items and is designed to evaluate a broad range of psychological problems and symptoms of psychopathology. It measures 9 primary symptom dimensions and is designed to provide an overview of a patient's symptoms and their intensity at a specific point in time.
Self-Esteem Scale | week 12 (end of treatment)
  Self-Esteem Scale (SES; Rosenberg, 1965; Polish version: Dzwonkowska, Lachowicz-Tabaczek & Łaguna, 2008). The SES is a 10-item self-report scale that measures global self-worth by measuring both positive and negative feelings about the self.
Defense Style Questionnaire | week 12 (end of treatment)
  Defense Style Questionnaire (DSQ-40; Andrews, Singh & Bond M, 1993; Polish version: Bogutyn, Kokoszka, Pałczyński & Holas, 1999). The DSQ-40 is a 40 item self-report questionnaire designed to measure an individual's propensity towards three various defense styles (mature, neurotic and immature) along with twenty individual defense mechanisms.
Personality Beliefs Questionnaire | week 12 (end of treatment)
  Personality Beliefs Questionnaire (PBQ; Beck & Beck, 1991; Polish translation). The PBQ is a 126-item self-report measure of beliefs associated with 10 DSM-III-R and DSM-IV personality disorders (represented as subscales): 1) avoidant; 2) dependent; 3) obsessive-compulsive; 4) histrionic; 5) passive-aggressive; 6) narcissistic; 7) paranoid; 8) schizoid; 9) antisocial, and 10) borderline.
Inventory of Interpersonal Problems | week 12 (end of treatment)
  Inventory of Interpersonal Problems (IIP; Horowitz, Alden, Wiggins, & Pincus 2000; Polish translation). The IIP is a 64-item self-report questionnaire that inventories the interpersonal problems that people experience. It contains eight scales that assess different aspects of an individual's interpersonal difficulties: 1) domineering/controlling; 2) vindictive/self-centered; 3) cold/distant; 4) socially inhibited; 5) non-assertive; 6) overly accommodating; 7) self-sacrificing; 8) intrusive/needy.
Dysfunctional Working Models Scale | week 12 (end of treatment)
  Dysfunctional Working Models Scale (DWM-S; Perris, Fowler, Skagerlind, Olsson & Thorsson, 1998; Polish version: Nieznański, Habrat, Szyszkowski, Chojnowska & Walczak, 2001). The DWM-S is a 35-item self-report measure of dysfunctional working models of self and others.
Experiences in Close Relationships | week 12 (end of treatment)
  Experiences in Close Relationships (ECR; Brennan , Clark & Shaver, 1998; Polish version: Stawska, 2010). The ECR is a 36-item self-report measure of adult attachment. It groups people into four different categories on the basis of scores along two scales: avoidance and anxiety.
Bell Object Relations and Reality Testing Inventory | week 12 (end of treatment)
  Bell Object Relations and Reality Testing Inventory (BORRTI; Bell, 1995; Polish version: Staniszewski, 2011). The BORRTI is a 45-item self-report measure designed to evaluate the ability to sustain essential relationships and accurately identify internal and external reality.
Meta-cognitions Questionnaire | week 12 (end of treatment)
  Meta-cognitions Questionnaire (MCQ; Cartwright-Hatton & Wells, 1997; Polish version: Gawęda & Kokoszka, 2013). The MCQ is a 65-item self-report scale developed to assess several dimensions of metacognition thought to be relevant to psychopathology. Its ﬁve subscales are: 1) positive beliefs about worry; 2) negative beliefs about thoughts concerning uncontrollability and danger; 3) cognitive conﬁdence (assessing conﬁdence in attention and memory); 4) negative beliefs concerning the consequences of not controlling thoughts, and 5) cognitive self-consciousness (the tendency to focus attention on thought processes).
Five Facet Mindfulness Questionnaire | week 12 (end of treatment)
  Five Facet Mindfulness Questionnaire (FFMQ-S; Baer et al. 2006; Polish translation). FFMQ-S is a 39-item self-report measure which assesses five facets of a general tendency to be mindful in daily life: observing, describing, acting with awareness, nonreactivity to inner experience, and nonjudging of inner experience.
Satisfaction With Life Scale | week 12 (end of treatment)
  Satisfaction With Life Scale (SWLS; Diener, Emmons, Larsen & Griffin, 1985; Polish version: Juczyński, 2001). The SWLS is a 5-item self-report global measure of life satisfaction.
Self-Esteem Scale | week 24 (follow-up)
  Self-Esteem Scale (SES; Rosenberg, 1965; Polish version: Dzwonkowska, Lachowicz-Tabaczek & Łaguna, 2008). The SES is a 10-item self-report scale that measures global self-worth by measuring both positive and negative feelings about the self.
Defense Style Questionnaire | week 24 (follow-up)
  Defense Style Questionnaire (DSQ-40; Andrews, Singh & Bond M, 1993; Polish version: Bogutyn, Kokoszka, Pałczyński & Holas, 1999). The DSQ-40 is a 40 item self-report questionnaire designed to measure an individual's propensity towards three various defense styles (mature, neurotic and immature) along with twenty individual defense mechanisms.
Personality Beliefs Questionnaire | week 24 (follow-up)
  Personality Beliefs Questionnaire (PBQ; Beck & Beck, 1991; Polish translation). The PBQ is a 126-item self-report measure of beliefs associated with 10 DSM-III-R and DSM-IV personality disorders (represented as subscales): 1) avoidant; 2) dependent; 3) obsessive-compulsive; 4) histrionic; 5) passive-aggressive; 6) narcissistic; 7) paranoid; 8) schizoid; 9) antisocial, and 10) borderline.
Inventory of Interpersonal Problems | week 24 (follow-up)
  Inventory of Interpersonal Problems (IIP; Horowitz, Alden, Wiggins, & Pincus 2000; Polish translation). The IIP is a 64-item self-report questionnaire that inventories the interpersonal problems that people experience. It contains eight scales that assess different aspects of an individual's interpersonal difficulties: 1) domineering/controlling; 2) vindictive/self-centered; 3) cold/distant; 4) socially inhibited; 5) non-assertive; 6) overly accommodating; 7) self-sacrificing; 8) intrusive/needy.
Dysfunctional Working Models Scale | week 24 (follow-up)
  Dysfunctional Working Models Scale (DWM-S; Perris, Fowler, Skagerlind, Olsson & Thorsson, 1998; Polish version: Nieznański, Habrat, Szyszkowski, Chojnowska & Walczak, 2001). The DWM-S is a 35-item self-report measure of dysfunctional working models of self and others.
Experiences in Close Relationships | week 24 (follow-up)
  Experiences in Close Relationships (ECR; Brennan , Clark & Shaver, 1998; Polish version: Stawska, 2010). The ECR is a 36-item self-report measure of adult attachment. It groups people into four different categories on the basis of scores along two scales: avoidance and anxiety.
Bell Object Relations and Reality Testing Inventory | week 24 (follow-up)
  Bell Object Relations and Reality Testing Inventory (BORRTI; Bell, 1995; Polish version: Staniszewski, 2011). The BORRTI is a 45-item self-report measure designed to evaluate the ability to sustain essential relationships and accurately identify internal and external reality.
Meta-cognitions Questionnaire | week 24 (follow-up)
  Meta-cognitions Questionnaire (MCQ; Cartwright-Hatton & Wells, 1997; Polish version: Gawęda & Kokoszka, 2013). The MCQ is a 65-item self-report scale developed to assess several dimensions of metacognition thought to be relevant to psychopathology. Its ﬁve subscales are: 1) positive beliefs about worry; 2) negative beliefs about thoughts concerning uncontrollability and danger; 3) cognitive conﬁdence (assessing conﬁdence in attention and memory); 4) negative beliefs concerning the consequences of not controlling thoughts, and 5) cognitive self-consciousness (the tendency to focus attention on thought processes).
Five Facet Mindfulness Questionnaire | week 24 (follow-up)
  Five Facet Mindfulness Questionnaire (FFMQ-S; Baer et al. 2006; Polish translation). FFMQ-S is a 39-item self-report measure which assesses five facets of a general tendency to be mindful in daily life: observing, describing, acting with awareness, nonreactivity to inner experience, and nonjudging of inner experience.
Satisfaction With Life Scale | week 24 (follow-up)
  Satisfaction With Life Scale (SWLS; Diener, Emmons, Larsen & Griffin, 1985; Polish version: Juczyński, 2001). The SWLS is a 5-item self-report global measure of life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Kokoszka, MD, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Hospital of Wola, Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Gibbon S, Khalifa NR, Cheung NH, Vollm BA, McCarthy L. Psychological interventions for antisocial personality disorder. Cochrane Database Syst Rev. 2020 Sep 3;9(9):CD007668. doi: 10.1002/14651858.CD007668.pub3. PMID 32880104
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Suszek H, Holas P, Wyrzykowski T, Lorentzen S, Kokoszka A. Short-term intensive psychodynamic group therapy versus cognitive-behavioral group therapy in day treatment of anxiety disorders and comorbid depressive or personality disorders: study protocol for a randomized controlled trial. Trials. 2015 Jul 29;16:319. doi: 10.1186/s13063-015-0827-6. PMID 26220089